CLINICAL TRIAL: NCT00431249
Title: Effects of Cilostazol on Vascular Endothelial Growth Factor , Inflammatory and Oxidative Stress Biomarkers in Hemodialysis Patients With Peripheral Vascular Disease.
Brief Title: Effects of Cilostazol on VEGF and Oxidative Stress Biomarkers in Hemodialysis Patients With Peripheral Vascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Principal Investigator, Paik Seong Lim, MD, Tungs' Taichung Metroharbour Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 960126
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Hemodialysis Patients; Peripheral Vascular Disease
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- one (Other)
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol

SUMMARY:
Peripheral arterial disease (PAD) is the most common manifestation of systemic atherosclerosis and accounts for significant morbidity and mortality among end-stage renal disease (ESRD) patients. However, few studies have identified the prevalence and clinical impact of PAD in this specific population.

Objectives: To perform a single-blinded parallel, controlled trial to examine the effect of cilostazol treatment on plasma VEGF levels, tissue factors , inflammatory markers (such as IL-6, hsCRP) levels, oxidative stress markers in ESRD patients with PAD Material and methods Fourty HD patients on maintenance HD for > 3months were enrolled in this prospective, single-blinded, randomized study. These patients were randomly allocated into 2 arms. After baseline assessment, patients in the treatment arm received 12 weeks of added on therapy with cilostazol 100mg/day. Blood pressure, heart rate, oxidative stress (malonyldialdehyde, protein carbonyl and ADMA), inflammatory markers (hsCRP, IL-6) and plasma, VEGF and tissue factors levels were measured before and after treatment.

DETAILED DESCRIPTION:
Purpose :

Patients with end stage renal disease are at an increased risk for cardiovascular disease (CVD) and the annual mortality from CVD in end-stage renal disease (ESRD) patients is substantially higher than in the general population. Peripheral arterial disease (PAD), the most common manifestation of atherosclerosis, is characterized by atherosclerotic occlusive disease of the lower extremities. The most common symptom of PAD is intermittent claudication, defined as pain, cramping, or aching in the calves, thighs, or buttocks. However, it has been reported that over one-half of those with PAD remains asymptomatic. Rest pain, tissue loss, and gangrene are among the more extreme presentations of PAD and PAD has been a major cause for lower-extremity amputation, especially in those HD patients with diabetes. However, few available data stressed on the huge burden of PAD in hemodialysis (HD) patients. More importantly, presence of PAD in these patients is an important predictor for subsequent cardiovascular and overall mortality. The medical therapy of in PAD in general population is limited to a few antiplatelet drugs and statin in relatively few descriptive studies and randomized control trials. There are no appropriate randomized trials of these therapies in the treatment of PAD in patients with chronic kidney diseases. Hence, there are as yet no substantial data to support for efficacy of pharmacologic interventions of PAD in these specific groups of patients.

Hypothesis

Use of cilosatzol may be associated with increased plasma levels of VEGF and TF and amelioration of inflammation in HD patients with PAD.to perform a parallel, controlled trial to examine the effect of cilostazol treatment on plasma VEGF levels, tissue factors , inflammatory markers (such as IL-6, hsCRP) levels, oxidative stress markers in ESRD patients with PAD.

Many human diseases are characterized by disorders of the vasculature. In ischemic heart disease or peripheral artery disease, insufficient blood vasculature leads to tissue ischemia. Out of the many players in the angiogenesis field, the vascular endothelial growth factors are by far the best characterized and several VEGFs have already entered clinical use in a variety of human conditions. While many studies have addressed the role of angiogenesis and the blood vasculature in human physiology and pathology, the role of proangiogenic therapy in PAD has until recently attracted very little attention. VEGF is the prime hypoxia inducible angiogenic factor and binds VEGFR-1 and VEGFR-2. VEGF increases permeability of the endothelium through the formation of intercellular gaps, vesico-vascular organelles, vacuoles as well as fenestrations. VEGF also causes vasodilatation through the induction of the endothelial nitric oxide synthase (eNOS) and the subsequent increase in nitric oxide production. In recent years, several studies have reported beneficial effects of VEGF when used as a proangiogenic therapy in the setting of tissue ischemia. While proangiogenic therapies could be employed in the treatment of various ischemic diseases,controlling these processes with targeted molecular therapies remains at the heart of research.

Cilostazol is a phosphodiesterase III inhibitor with a profound pharmacological profile. Cilostazol, {6[4-(1-cyclohexyl-1H-tetrazol-5-yl) butoxy]-3,4-dihydro-2-(1H)- quinolinone} is a 2-oxoquinolone derivative (molecular weight, 369.47) that has a plasma half-life of 10.564.4 hours after oral administration. It inhibits both primary and secondary platelet aggregation in response to ADP, collagen, epinephrine, and arachidonic acid. The antiplatelet and vasodilator properties of cilostazol have been attributed to its ability to elevate intracellular levels of cAMP.3 Cilostazol is currently used for treatment of symptomatic intermittent claudication (IC).Studies performed in diabetic patients have indicated that, in addition to its vasodilator and antiplatelet properties. Cilostazol may also favorably modify plasma lipoproteins by increasing HDL cholesterol (HDL-C) and reducing triglycerides. Numerous trials have evaluated the anti-proliferative properties of cilostazol and most found that it can prevent restenosis in patients undergoing percutaneous coronary intervention (PCI). In Japanese patients with type 2 diabetes, cilostazol therapy was associated with regression of carotid intimal thickness.

The observed efficacy of cilostazol is not fully explained. Most investigators hypothesized that cilostazol exhibits its pharmacologic effects via antiplatelet, vasodilatory, and antithrombotic activities. Other postulated mechanisms of cilostazol action include a) anti-proliferative function by preventing restenosis after PCI, b) improved lipid profiles and c) prevent atherosclerosis via inhibition of the expression of the adhesion molecule. Some of these hypotheses may be valid, but clearly more confirmatory studies are needed. Although cilostazol has all the above properties, its effect on the expression of VEGF and oxidative stress biomarkers is not known For that purpose, we plan to study the changes in lipoprotein levels, proangiogenetic factors, inflammation, oxidative stress and endothelial activation following 12 weeks of cilostazol in a group of 40 HD patients. We feel that the present study may help to shed some lights and broaden our understanding of the pathophysiological mechanisms underlying the beneficial effects of cilostazol and give further insights on the role of antiplatelet drugs in PAD both by improving clinical symptoms and plausibly by reducing cardiovascular events

ELIGIBILITY:
Inclusion Criteria:

1. Both sexes aged between 30-70 years
2. Non-diabetic ESRD Patients on HD greater than 3 months
3. Patients with PAD diagnosed by clinical symptoms, and ABI indices < 0.9 and confirmed by angiographic or related studies.
4. Written informed consent

Exclusion Criteria:

1. Known allergy to cilostazol
2. Patients who currently have had pentoxyphylline or related therapy
3. Congestive heart failure or cardiac arrhythmia
4. Severe liver impairment
5. Patients with malignancy or acute/chronic inflammatory diseases
6. Smoking during the previous 6 months
7. Recent stroke
8. Severe dyslipidemia (triglycerides >600 mg/dL or total cholesterol >300g/dL) or currently on statin therapy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Effects on Biomarkers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Palk Seong Lim, MD, Principal Investigator — Tungs' Taichung Metroharbour Hospital